CLINICAL TRIAL: NCT02597725
Title: Changes in Bladder Function After Surgery and Radiation Therapy for Prostate Cancer
Brief Title: Salvage Radiotherapy After Radical Prostatectomy
Acronym: SRT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Urodynamics in prostate cancer
Record Dates: First submitted 2015-10-07; First posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: Urodynamics; Late effects; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Urodynamics: There is no intervention in this study.

SUMMARY:
The purpose of this study is to describe the urinary morbidity as a result surgery and radiation therapy, in patients treated for prostate cancer.

All the patients will undergo a Urodynamic examination to verify the grade of Urinary morbidity.

DETAILED DESCRIPTION:
Introduction:

There is a little knowledge on long-term urinary morbidity in patients treated with radical prostatectomy (RP) and salvage radiotherapy (SRT). Both treatments are potentially curative for localized prostate cancer (PC). Improved long-term survival makes the awareness of late effects from radiotherapy important.

Purpose:

The purpose of this study was to access, late urinary morbidity in patients treated with SRT. The patients included in this study will have an urodynamic examination. The results from the urodynamic examination will help us with a better understanding of the different symptoms and their grade, after treatment with RP and SRT because of PC.

Materials and methods:

A total of 67 patients will be invited to participate in this urodynamic study. The patients will undergo a urodynamic examination, included biomechanical examination of urethra. The examination is a standard procedure at the department of Urology, Aarhus University hospital, Denmark.

The patients will, in relation to the urodynamics, have taken two blood samples. The blood samples, will later on, be used to detect some of the genetic reasons for morbidity after radiotherapy.

Endpoint:

The primary endpoint is the outcome of different parameters as a result of the urodynamic examination.

Perspective:

The perspective of this study is to help understanding the efficacy og morbidity of salvage radiotherapy. The investigators hope to get a better understanding of the mechanisms related to urinary morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with salvage radiotherapy at Aarhus University hospital in the period from 2006-2010.

Exclusion Criteria:

* Other cancer types
* Severe comorbidity

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in this cohort had surgery for prostate cancer in the period from 1999-2009. Because of a locale disease relapse the patients were treated with Salvage radiation therapy in the period from 2006-2010.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Spontaneous urinary flow | 2 minutes
  The patients load the water at a special flow toilet
Biomechanical properties of urethra | 10 minutes
  Evaluation of biomechanical wall properties by measuring luminal cross-sectional area and pressure.
Cystometri | 20 minutes
  The bladder is filled with saline with a flow rate of 60 mL/minute.
Uretal pressure profile | 10 minutes
  To evaluate the uretal pressure profile. The water pump perfused saline at a flow rate of 1 mL, while the catheter. attached to an automatic pulling device, was pulled out of the urethra at 2 mm/s.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borre, Professor, Study Chair — University of Aarhus; Morten Høyer, Professor, Study Chair — University of Aarhus